CLINICAL TRIAL: NCT01133652
Title: The VISION STUDY: Variation In Success of Intravenous (IV) Placement With Observation Using New Techniques
Brief Title: Variation In Success of Intravenous (IV) Placement With Observation Using New Techniques
Acronym: VISION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Sarah Curtis, Dr. Sarah Curtis, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00004389; G049000062 (Other Grant/Funding Number: Womens and Children's Health Research Institute)
Record Dates: First submitted 2010-05-18; First posted 2010-05-31 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Catheterization; Peripheral Phlebotomy
Keywords: Venipuncture; Randomized Controlled Trial; Intravenous access; Children; Pediatric Emergency Department; Peripheral intravenous catheterization; Catheterization, Peripheral Phlebotomy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- VeinViewer (Active Comparator): The Veinviewer machine will be used to guide intravenous access.
  Interventions: Device: Veinviewer
- Ultrasound (Active Comparator): The Ultrasound will be used to guide intravenous access.
  Interventions: Device: Ultrasound
- Conventional IV placement (Active Comparator): IV will be placed using conventional technique
  Interventions: Other: Conventional technique

INTERVENTIONS:
Device: Veinviewer — Veinviewer machine
  Arms: VeinViewer
Device: Ultrasound — Ultrasound
  Arms: Ultrasound
Other: Conventional technique — Conventional IV placement by nurses
  Arms: Conventional IV placement

SUMMARY:
Children fear having an intravenous (IV) needle placed because of the pain that they will experience. The more needle punctures that a child has to endure before the IV is successfully placed, the greater the pain experienced and anxiety suffered. In addition, false starts increase the demands on medical staff and can increase the length of the emergency department stay. Often, veins are difficult to see or feel, particularly in an unwell, dehydrated child or in young infants who have more fat below the skin surface. Also, the venous pattern below the skin surface naturally varies from person to person and therefore success in placing IVs leaves room for improvement. Technology may be able to play an important role is improving the rates of success. The investigators wish to investigate whether the use of either an Ultrasound machine or a VeinViewer machine can improve the rate of success of the initial attempt (skin puncture) at peripheral IV placement in comparison to the current standard approach.

DETAILED DESCRIPTION:
Peripheral IV line placement is one of the most common and challenging painful procedures performed in the pediatric emergency department (PED). The lack of a clear visual guide for IV placement often leads to multiple painful attempts; delays in urgent treatment; increased use of human resources; increased costs; and increased anxiety in the patient, the parents and the staff. The research plan is a randomized controlled trial (RCT) to compare the use of two new technologies with the current standard method for vein location and IV placement in children.We would like to know if either of these technologies improve rates of successful IV placement on first attempt. Furthermore we would like to know if either technology leads to decreased time spent by staff on the procedure or decreased overall number of painful attempts. Information on nursing satisfaction, parental satisfaction and cost analysis will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-16 presenting to the Pediatric Emergency Department (PED)
* Require IV as part of routine care
* Knowledge of English language

Exclusion Criteria:

* Child in critical condition
* Child requires urgent IV placement
* Central line available

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 399 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Success or failure of peripheral IV placement on first attempt. | Within one hour of start of procedure
  The time to placement of a successful intravenous catheter is variable but is generally completed within one hour. This is an estimated timeframe.

SECONDARY OUTCOMES:
Number of attempts to successful IV placement | Within one hour of start of procedure
  The time to placement of a successful intravenous catheter is variable but is generally completed within one hour. This is an estimated timeframe.
Time to successful placement of IV | Within one hour
  The time to placement of a successful intravenous catheter is variable but is generally completed within one hour. This is an estimated timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Curtis, MD, Principal Investigator — Division of Pediatric Emergency Medicine, Department of Pediatrics & Women and Children's Health Research Institute
Locations (1):
- Stollery Children's Hospital Pediatric Emergency Department, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Curtis SJ, Craig WR, Logue E, Vandermeer B, Hanson A, Klassen T. Ultrasound or near-infrared vascular imaging to guide peripheral intravenous catheterization in children: a pragmatic randomized controlled trial. CMAJ. 2015 May 19;187(8):563-570. doi: 10.1503/cmaj.141012. Epub 2015 Apr 20. PMID 25897047